CLINICAL TRIAL: NCT05123781
Title: An Open, Comparative, Randomized, Crossover, Bioequivalence Study of Metformin, Prolonged-release Tablets 500 mg (JSC Farmak, Ukraine) vs Glucophage® XR in Healthy, Adult Male and Female Subjects Under Fasting Conditions
Brief Title: Fasting Bioequivalence Study of 2 Metformin 1000 mg Prolonged Release Tablets in 28 Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/MTF/FS
Record Dates: First submitted 2021-11-09; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Metformin 1000 mg Prolonged Release Tablets; Prolonged Release Tablets; oral dosage form; Metformin
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine)
  Interventions: Drug: Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine)
- Treatment B (Active Comparator): Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK)
  Interventions: Drug: Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK)

INTERVENTIONS:
Drug: Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) — One tablet of the test product was administered orally with 240 ml of water
  Other Names: Diaformin® SR 1000mg tablets (JSC Farmak, Ukraine); Diabufor® XR 1000mg tablets (JSC Farmak, Ukraine)
  Arms: Treatment A
Drug: Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK) — One tablet of the Reference product was administered orally with 240 ml of water
  Other Names: Glucophage® XR 1000 mg
  Arms: Treatment B

SUMMARY:
The primary objective was to compare the rate and extent of absorption of Metformin XR after administration of a Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK), administered as a single dose in healthy subjects under fasting conditions.

The adverse events, physical examinations and vital signs were reported for the evaluation of safety.

DETAILED DESCRIPTION:
An Open, Comparative, Randomized, Crossover Clinical Trial to Evaluate the Bioequivalence of Single Doses of Test Product Metformin 1000 mg Prolonged Release Tablets (JSC Farmak, Ukraine) and Reference Product Glucophage® XR 1000 mg Prolonged Release Tablets (Merck Serono Ltd, UK) in Healthy, Adult Male and Female Subjects Under Fasting Conditions.

Single oral dose of Test of Reference product of Metformin 1000 mg Prolonged Release Tablets was administered to volunteers under fasting conditions in the morning of Day 1 of each Study Period.

The study consists of two study periods with a washout period of at least 7 days between doses.

During each study period 21 blood samples were taken: prior to dosing (-1.0) and 1.0, 2.0, 3.0, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 8.5, 9.0, 10.0, 12.0, 16.0, 24.0, 32.0 and 36.0 hours after IMP administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and non-pregnant and no breast-feeding females (must have a negative pregnancy test result prior to dosing). Caucasian race.
2. Non-smoker or past-smoker (who has stopped smoking at least 6 months before the first dosing).
3. Body Mass Index (BMI) 18.5 to 30.0 kg/m2, inclusive and body weight between 50 kg and 100 kg (on the day of screening).
4. Subject is available for the whole study and has provided his/her written informed consent.
5. Subjects in good health, as determined by screening medical history, physical examination, vital signs assessments (pulse rate, systolic and diastolic blood pressure, and body temperature) and 12-lead ECG. Minor deviations outside the reference ranges will be acceptable, if deemed not clinically significant by the Investigator.
6. Subjects in good health and with glucose between 3.3 mmol/L-5.5 mmol/l at screening, as determined by screening clinical laboratory evaluations. Minor deviations outside the reference ranges will be acceptable, if deemed not clinically significant by the Investigator. 7. Acceptance of use of contraceptive measures during the whole study by both female and male subjects

Exclusion Criteria:

1. Known cardiovascular disease, history of hypotension.
2. Factors in the subject's history that may predispose to ketoacidosis and lactic acidosis or all types of the metabolic acidosis (including pancreatic insulin deficiency, history of pancreatitis, caloric restriction disorders, restricted food intake, alcohol abuse)
3. Gastrointestinal, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
4. Previous liver disease or elevations in serum transaminases ALT or AST ≥1.0 ULN at the screening (for women 0-0.52 µmol/L and for men 0-0.68 µmol/L).
5. Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the IMP.
6. History of kidney disease with impaired renal function and level of creatinine out of the normal laboratory range based on screening.
7. History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs.
8. Clinically significant illness within 28 days before the first dosing, including major surgery.
9. Any significant clinical abnormality, including a positive result of HBsAg and/or HCV and/or HIV test during screening procedure.
10. Positive screening urine drugs abuse test or/and alcohol breath test or urine cotinine test, and positive pregnancy test on screening.
11. Serious mental disease and/or inability to cooperate with clinical team.
12. Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 100-140 mmHg for systolic BP and/or 60-100 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
13. Body ear temperature is out of the range of 35.7-37.6°C at screening.
14. Orthostatic hypotension during the screening procedure.
15. Drug, alcohol (of ≥ 40 g per day pure ethanol), solvents or caffeine abuse.
16. Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 90 days before the first dosing.
17. Use of any prescription medication for a period of 28 days before the first dosing.
18. Any systemic over-the-counter (OTC) drug treatment and/or vitamins and/or herbal treatment/or food supplements within 14 days before the first dosing.
19. Getting a tattoo, body piercing or any cosmetic treatment involving skin piercing within 90 days before the screening unless evaluated by Investigator as non-significant for inclusion in the study.
20. Donation or loss of at least 500 mL of blood within 90 days or donation of plasma or platelets within 14 days before the first dosing.
21. Anaemia, haemoglobin below 120 g/L for women and 130 g/L for men at screening. 22. Less than 30 days between exit procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to 36 hours post-administration
  area under the plasma drug concentration
Cmax | up to 36 hours post-administration
  maximum plasma concentration observed.

SECONDARY OUTCOMES:
AUC(0-∞) | up to 36 hours post-administration
  area under the plasma drug concentration versus time curve from time zero to infinity
AUC(0-12h) | from time zero to time 12 hours after dosing
  the area under the plasma drug concentration versus time curve calculated from time zero to time 12 hours after dosing
AUC(12h-t) | from time 12 hours after dosing to time of the last sample above LLOQ.
  the area under the plasma drug concentration versus time curve calculated from time 12 hours after dosing to time of the last sample above LLOQ.
AUC(0-24h) | from time zero to time 24 hours after dosing
  the area under the plasma drug concentration versus time curve calculated from time zero to time 24 hours after dosing.
tmax | up to 36 hours post-administration
  the time of the maximum plasma drug concentration.
λz | up to 36 hours post-administration
  apparent first-order elimination
t1/2 | up to 36 hours post-administration
  the elimination or terminal half-life
AUCres | up to 36 hours post-administration
  Residual area

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- QUINTA-ANALYTICA s.r.o., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No